CLINICAL TRIAL: NCT03915665
Title: Non-surgical Treatment of Peri-implant Mucositis: A Randomized Controlled Clinical Trial Comparing Standard Treatment and Comprehensive Treatment
Brief Title: Non-surgical Treatment of Peri-implant Mucositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NSTPM
Record Dates: First submitted 2018-12-30; First posted 2019-04-16 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Peri-implant Mucositis
MeSH Terms: interventions — Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment (Active Comparator): Manual treatment One application of Chlorhexidine 1% gel
  Interventions: Drug: Chlorhexidine
- Comprehensive treatment (Experimental): Supragingival biofilm removal with Erythritol air-powder Submucosal biofilm removal with Erythritol air-powder (30%-60% power)
  Interventions: Device: Air-powder

INTERVENTIONS:
Drug: Chlorhexidine — Chlorhexidine gel 1% one single application after mechanical biofilm removal through manual instruments
  Arms: Standard treatment
Device: Air-powder — Erythritol powder using air-powder device
  Arms: Comprehensive treatment

SUMMARY:
This a Randomized Controlled Clinical Trial comparing two techniques for the nonsurgical treatment of peri-implant mucositis. The main objective of the present randomized controlled clinical trial is to determine whether the application of a novel treatment strategy for peri-implant mucositis could lead to significantly improved clinical parameters as compared to standard treatment. Half of the patients receives treatment with manual instruments and chlorhexidine gel 1%, half receives treatment with submucosal biofilm removal by erythritol powder.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should have at least one implant (Renvert et al. 2009),
* with bleeding on probing using a 0.2N probing force or spontaneous bleeding with local swelling (code 1, 2 or 3 as described in Corbella et al. 2011) and with bone resorption of no more of 1 mm (preferably no bone loss visible on radiographs) as evaluated through the use of standardized radiographs, taken with the use of an individualized radiograph holder in comparison with findings from radiographs taken immediately following placement of the implant prosthesis (similar to Renvert et al. 2009 and Algraffee et al. 2011).
* females and males 35 to 65 years old; (IV) full mouth bleeding score % lower than 20%.

Exclusion Criteria:

* systemic diseases that could affect the immune response or that could condition the bacterial colonization
* use of anti-inflammatory prescription medications, or antibiotics within the preceding respectively 1 week and 3 months or during the study,
* full-mouth plaque score (FMPS) >20%;
* full-mouth bleeding score (FMBS) >20%,
* smokers of more than 5 cigarettes a day,
* Documented allergy or intolerance towards the components of the products used in the study,
* Presence of active infection with suppuration.
* Absence of periodontitis in the rest of the mouth
* Pregnancy (certified by auto-declaration)
* Patients suffering from upper respiratory tract infections, from chronic bronchitis
* endocarditis, breast feeding, contagious disease, immune deficiency (neutropenia, angranulocytosis, diabetes, hemophilia), patients under treatment (radiotherapy, chemotherapy, antibiotics).

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
Bleeding index change | 3 months
  The primary outcome measure is the change in bleeding index between the baseline and the follow-up visit, on the basis of the following index: 0) no bleeding; 1) bleeding on probing without redness and swelling; 2) bleeding on probing, redness and swelling; and 3) spontaneous bleeding.

SECONDARY OUTCOMES:
PPD changes | 2 weeks, 1 month, 3, 6, 12, 24 months
  Changes in peri-implant probing depth between baseline and follow-up visit
Tissue level changes | 2 weeks, 1 month, 3, 6, 12, 24 months
  Changes in tissue level between baseline and follow-up visit, measured as the distance between a reference point on an occlusal personalized stent, made with polyvinylsiloxane impression material, and the mucosal margin
PI changes | 2 weeks, 1 month, 3, 6, 12, 24 months
  Changes in plaque index between baseline and follow-up visit on the basis of the following indeX: 0) no plaque accumulation; 1) plaque accumulation only detectable using a probe; 2) moderate accumulation of visible plaque/ calculus; 3) high accumulation of visible plaque/calculus.)
BI changes | 2 weeks, 1 month, 6, 12, 24 months
  The primary outcome measure is the change in bleeding index between the baseline and the follow-up visit, on the basis of the following index: 0) no bleeding; 1) bleeding on probing without redness and swelling; 2) bleeding on probing, redness and swelling; and 3) spontaneous bleeding.
Marginal bone level changes | 6 and 12 months
  Changes in radiographic marginal bone level between baseline and follow-up visit measured comparing the periapical radiograph (with individualized holder) taken during baseline visit and the ones taken 6 and 12 months after intervention.
Pain perception: Visual Analogue Scale | Immediately after intervention
  Pain perception during intervention, measured with a 10-mm long Visual Analogue Scale scale being 0 equal to no pain and 10 equal to maximum, unbearable, pain. Lower values represent better outcome.
Limitations in daily activity | 7 days
  Limitations in daily activity measured with a 10-mm long VAS scale being 0 equal to no limitation and 10 equal to complete limitation in daily activity, recorded daily. Lower values represent better outcome.
Taste alteration | 7 days
  Alteration in taste measured with a 10-mm long VAS scale being 0 equal to no alteration and 10 equal to complete taste alteration, recorded daily. Lower values represent better outcome.
Taste sensation | 7 days
  Taste sensation measured with a 10-mm long VAS scale being 0 equal to no sensation and 10 equal to revolting taste sensation, recorded daily. Lower values represent better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided
The investigators planned to share anonymized IPD after the end of the study